CLINICAL TRIAL: NCT04118140
Title: Development and Preliminary Evaluation of an Evidence-based Somatic Acupressure Protocol for the Self-management of Symptom Cluster of Fatigue, Insomnia and Depression in Breast Cancer Patients
Brief Title: Somatic Acupressure for Symptom Cluster Management in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H19017
Record Dates: First submitted 2019-09-27; First posted 2019-10-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Cancer
Keywords: Cancer; acupressure; fatigue; depression; insomnia; symptom cluster
MeSH Terms: conditions — Neoplasms; Fatigue; Depression; Sleep Initiation and Maintenance Disorders; Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study can perform a partial blind design for participants in the true and sham intervention groups. Blind of outcome assessment will be also achieved in the true and sham intervention groups as all the questionnaires are patient-reported and the participants themselves will be the outcome assessors. Data analysis will be conducted by an independent statistician who are blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True SA (Somatic Acupressure ) group (Experimental): Receiving true somatic acupressure+usual care
  Interventions: Other: Somatic Acupressure; Other: Usual care
- Sham SA group (Sham Comparator): Receiving sham somatic acupressure+usual care
  Interventions: Other: Sham acupressure; Other: Usual care
- Usual care group (Other): Receiving usual care only (an education booklet regarding knowledge of BC and FSD symptom cluster management advice)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Somatic Acupressure — 7-week self-acupressure plus usual care (an education booklet)
  Arms: True SA (Somatic Acupressure ) group
Other: Sham acupressure — Same dose as the true acupressure group but on the sham acupoints plus usual care (an education booklet)
  Arms: Sham SA group
Other: Usual care — Usual care only (an education booklet)

SUMMARY:
Using a robust research method following the MRC Framework, the proposed study will develop and test an evidence-based complementary health intervention to help breast cancer patients manage the fatigue-sleep disturbance-depression symptom cluster.

DETAILED DESCRIPTION:
The fatigue-sleep disturbance-depression (FSD) symptom cluster is one of the most common symptom clusters in breast cancer (BC) patients, which can significantly deteriorate patients' functional status and quality of life. Since symptom cluster management has been unsatisfactory by using pharmacological treatments alone, the use of non-pharmacological adjuvant approaches has therefore been recommended. Being an important modality of acupoint stimulation, somatic acupressure (SA) can be a promising non-pharmacological intervention given its potential benefits for cancer symptom alleviation and its convenience for self-practice without increasing patients' physical and financial burden. However, current research on acupoint stimulation for cancer symptom management has been mainly focusing on individual symptom, and intervention protocols have been found significantly varied in intervention dosages and acupoint formula without a standardised protocol developed via a rigorous evidence-based research approach. The proposed study therefore follows the Medical Research Council (MRC) Framework for Developing and Evaluating Complex Intervention (the MRC Framework) to develop an evidence-based SA protocol to help with a better management of the FSD symptom cluster in BC. The first two phases of the MRC Framework will be included in this study. The first phase utilizes an evidence-based method to comprehensively review all available research evidence on acupoint-stimulation for cancer-related fatigue, sleep disturbance and depression, and further identify the most effective acupoint formula with the optimal SA duration and frequency. A preliminary SA protocol will then be developed based on the current research evidence and relevant theories and guidelines of acupoint stimulation. A content validity study will be conducted then to examine the content validity of the SA protocol via an expert panel. In the second phase, a feasibility randomized controlled trial (RCT) will be conducted to examine the acceptability of the SA protocol, pilot the methodological procedure of the clinical trial and preliminarily examine the effects of SA on the FSD symptom cluster in BC. Semi-structured interviews will be conducted afterwards to explore patients' experiences of participating in the study and receiving the SA.

ELIGIBILITY:
Inclusion Criteria:

1. BC stage I to IIIa;
2. have experienced at least a moderate level of the FSD symptom cluster, with a score of 4 or above on a 10-point numeric rating scale, from "0 (no symptom)" to "10 (worst symptom)", for each symptom during the past one month;
3. have completed adjuvant chemotherapy for at least one month and up to three years;
4. have not scheduled chemotherapy and radiotherapy during the whole study period;
5. willing to participate in the RCT and provide written informed consent.

Exclusion criteria:

1. presently taking pharmaceutical agents to treat fatigue, sleep disturbance or depression, such as antidepressant medications, psychostimulants, or hypnotics;
2. extremely weak and/or have cognitive impairment which make them unable (or difficult) to follow the study procedures and instructions;
3. having the experience of any types of SAS treatment during the past six months;
4. presently participating in any other research projects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
FEASIBILITY: Eligibility rate | Immediately after completion of the intervention (T2)
  Eligibility rate as assessed by (the number of eligible participants / number of participants screened) x 100%
FEASIBILITY: Recruitment rate | Immediately after completion of the intervention (T2)
  Recruitment rate as assessed by (the number of participants who participated in the study / number of eligible participants) x 100%
FEASIBILITY: Retention rate | Immediately after completion of the intervention (T2)
  Retention rate as assessed by (the number of participants who completed the study / number of participants who enrolled in) x 100%
FEASIBILITY: Attrition rate | Immediately after completion of the intervention (T2)
  Attrition rate as assessed by (the number of participants who dropped out after the randomization / number of participants who enrolled in) x 100%
FEASIBILITY: subject recruitment | Immediately after completion of the intervention (T2)
  Feasibility of subject recruitment assessed by interviewing the participants' feedback regarding why they discontinued this study
FEASIBILITY: Duration for completing the subject recruitment | Immediately after completion of the intervention (T2)
  Time period from the recruitment of first participants to the last patient: assessed by months
ACCEPTABILITY: Actual days of acupressure | Immediately after completion of the intervention (T2)
  The number of days that the participants perform the SA interventions, where the scheduled sessions should be 7 weeks of daily acupressure
ACCEPTABILITY: duration of each acupressure session | Immediately after completion of the intervention (T2)
  Duration of each time (minutes) of acupressure where the scheduled time per session should be around 36 minutes
ACCEPTABILITY: SA protocol | Immediately after completion of the intervention (T2)
  Participants' feedback and satisfaction with the SA intervention assessed by a self-designed feedback form and follow-up semi-structured interviews
FEASIBILITY: Questionnaire-Item-level missing value of each questionnaire | Immediately after completion of the intervention (T2)
  Item-level missing value of each questionnaire (%) assessed by the percentage of participants who do not answer any single item
FEASIBILITY: Questionnaire-Scale-level missing value of the questionnaire | Immediately after completion of the intervention (T2)
  Scale-level missing value of the questionnaire (%) assessed by the percentage of participants who do not answer at least one item in the whole questionnaire
SAFETY: adverse events | Immediately once an adverse event occurs
  Number of adverse events occur during the intervention

SECONDARY OUTCOMES:
Fatigue | Data collection will be conducted at baseline (T1) and immediately after completion of the intervention (T2)
  Fatigue measured by the Multidimensional Fatigue Inventory
Sleep disturbance | Data collection will be conducted at baseline (T1) and immediately after completion of the intervention (T2)
  Insomnia measured by Pittsburgh Sleep Quality Index
Depression | Data collection will be conducted at baseline (T1) and immediately after completion of the intervention (T2)
  Depression measured by Hospital Anxiety and Depression Scale
Patients' quality of Life | Data collection will be conducted at baseline (T1) and immediately after completion of the intervention (T2)
  Measured by the Functional Assessment of Cancer Therapy-Breast Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yu (Benjamin) Tan, PhD RN, Principal Investigator — Charles Darwin University
Locations (1):
- The Affiliated Hospital Of Southwest Medical University, Luzhou, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang T, Tan JB, Liu XL, Zheng SL, Zhao I, Eliseeva S, Polotan MJ, Cheng HL, Huang HQ. Implementing an evidence-based somatic acupressure intervention in breast cancer survivors with the symptom cluster of fatigue, sleep disturbance and depression: study protocol of a phase II randomised controlled trial. BMJ Open. 2022 Jan 20;12(1):e054597. doi: 10.1136/bmjopen-2021-054597. PMID 35058263